CLINICAL TRIAL: NCT01232153
Title: Preoxygenation Before Prehospital Tracheal Intubation With NIV Versus Balloon. A Multicenter Randomized Controlled Trial in Mobile Medical Emergency Rescue Service
Brief Title: Preoxygenation Before Prehospital Tracheal Intubation With NIV Versus Balloon
Acronym: PREOXY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: departure without replacement of the principal investigator
Sponsor: Hopital of Melun (Other)
Collaborators: Service d'Aide Médicale Urgente de Seine et Marne (Unknown)
Responsible Party: Principal Investigator, Sebastien Jochmans, MD, MD, Hopital of Melun
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PREOXY
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Preoxygenation
Keywords: chest tube; preoxygenation; NIV; out-of-hospital; patients needing tracheal chest tube managed by Medical Mobile Emergency rescue services
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIV preoxygenation (Active Comparator)
  Interventions: Device: Non invasive ventilation
- Classical preoxygenation (No Intervention)

INTERVENTIONS:
Device: Non invasive ventilation — Non invasive ventilation
  Arms: NIV preoxygenation

SUMMARY:
Recent studies reports feasibility, effectiveness and even less complications of using NIV for preoxygenation during tracheal intubation in ICU and in Operating Room. None study has been done in emergency out-of-hospital medical rescue. This trial attempts to demonstrate same results or even more in that conditions.

DETAILED DESCRIPTION:
This trial will compare classical preoxygenation strategy with unidirectional valve autofilling balloon versus NIV.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing chest tube intubation

Exclusion Criteria:

* Cardiac arrest
* Children
* Pregnancy
* Incompetents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
length of hypoxemia | 5 minutes
  SpO2 below 85%

CONTACTS AND LOCATIONS:
Locations (1):
- SAMU 77, Melun, France

IPD SHARING:
Plan to Share IPD: Undecided